CLINICAL TRIAL: NCT05921253
Title: Neuromodulation of Cardiovascular Risks Associated With Cardiotoxic Chemotherapy: A First in Human Randomized Pilot Study. Neuromodulation in Cancer Study (OU-SCC-NCAN)
Brief Title: Neuromodulation of Cardiovascular Risks Associated With Cardiotoxic Chemotherapy
Acronym: OU-SCC-NCAN
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Device Feasibility
Other Study IDs: OU-SCC-NCAN
Record Dates: First submitted 2023-06-12; First posted 2023-06-27 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Lymphoma
Keywords: Stimulation Device; Vagus Nerve Stimulator
MeSH Terms: conditions — Breast Neoplasms; Lymphoma

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, sham controlled, double-blinded study of low-level tragus stimulation vs. sham treatment.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Self administration of Low Level Tragus Stimulation (LLTS; Placebo) (Placebo Comparator): PARASYM neuromodulation device will be placed in a pre-determined position of one ear for 1 hour every day for 14 days.
  Interventions: Device: PARASYM neuromodulation device
- Self administration of LLTS (Experimental): PARASYM neuromodulation device will be placed in a pre-determined position (different from that of the placebo) of one ear for 1 hour every day for 14 days.
  Interventions: Device: PARASYM neuromodulation device

INTERVENTIONS:
Device: PARASYM neuromodulation device — Patients with breast cancer or lymphoma who have undergone chemotherapy for their disease, will have tests to determine heart function. Patients will be asked to use a handheld electrical unit (stimulator) at home to deliver vagus nerve stimulation (low level stimulation) to a preset position of one ear for a period of 1 hour for 14 days. After approximately 14 days, patients will have the same tests that they had at the beginning of the study.
  Other Names: Experimental
  Arms: Self administration of LLTS
Device: PARASYM neuromodulation device — Patients with breast cancer or lymphoma who have undergone chemotherapy for their disease, will have tests to determine heart function. Patients will be asked to use a handheld electrical unit (stimulator) at home to deliver vagus nerve stimulation (low level stimulation) to a different position of one ear compared to the "experimental arm" for a period of 1 hour for 14 days. After approximately 14 days, patients will have the same tests that they had at the beginning of the study.
  Other Names: Placebo
  Arms: Self administration of Low Level Tragus Stimulation (LLTS; Placebo)

SUMMARY:
This study is to determine if low level vagus nerve stimulation will lead to improvement in heart function, heart rate variation, and in the levels of certain chemical markers of inflammation in study participants' blood.

DETAILED DESCRIPTION:
Patients will be asked to use a handheld electrical unit (stimulator) at home to deliver vagus nerve stimulation (low level stimulation) to one ear for a period of 1 hour for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients (>18 years) who have received anthracycline-based therapy for breast cancer or lymphoma within the last 30 days
* A least 1 of following additional criteria:

  * previous chest radiation

    . Age>50
  * type 2 diabetes mellitus
  * hypertension
  * current smoking
  * obesity (BMI ≥ 30)
  * previous myocardial infarction
  * established atherosclerotic heart disease or significant valve disease. chronic kidney disease

Exclusion Criteria:

* Atrial paced rhythm
* History of seizure currently on treatment
* History of vasovagal syncope
* End stage liver or kidney disease

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Effects of low-level tragus stimulation (LLTS) on global longitudinal strain (GLS) | 2 weeks
  An echocardiogram will be performed on patients at baseline and at follow up (14 days after start of intervention). The percentage change of GLS and left ventricular ejection fraction (LVEF) will be compared at baseline and follow up in patients receiving cardiotoxic chemotherapy.

SECONDARY OUTCOMES:
Effects of LLTS on autonomic tone | 2 weeks
  Measure change in autonomic tone by 15-minute Heart Rate Variability at baseline and follow up. (2 week) HRV has time and frequency domain numbers that are continuous variables from 0-100 and more.
Effects of LLTS on oxidative stress | 2 weeks
  Analyze markers of oxidative stress in serum collected from patients at baseline and at follow up. Serum will be analyzed for oxidative stress before and after use of the TENS device. Results are expressed in Units - continuous variable.

CONTACTS AND LOCATIONS:
Overall Officials: Tarun W. Dasari, MD, MPH, Principal Investigator — University of Oklahoma
Locations (2):
- United States (2):
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Stephenson Cancer Center- Tulsa, Tulsa, Oklahoma

IPD SHARING:
Plan to Share IPD: No